CLINICAL TRIAL: NCT00189527
Title: Assist Control Versus Pressure Support Modes for Domiciliary Noninvasive Ventilation
Brief Title: Assist Control Versus Pressure Support Modes for Domiciliary Noninvasive Ventilation in Chronic Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche (Other)
Responsible Party: Pr A Cuvelier, CHU Rouen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2000-2
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Chronic Respiratory Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- respiratory support (Experimental): a mode of ventilation in comparison
  Interventions: Procedure: respiratory settings
- Assist Control (Active Comparator): an other mode of ventilation in comparison
  Interventions: Procedure: respiratory settings

INTERVENTIONS:
Procedure: respiratory settings

SUMMARY:
Noninvasive ventilation is a therapeutic option in some patients with chronic respiratory failure. Patients usually ventilate during nightime with a domiciliary ventilator either in assist control or in pressure support mode.

The aim of this study is to compare the clinical efficacy and the tolerance of assist control and pressure support modes during domiciliary noninvasive ventilation in patients with chronic respiratory failure.

DETAILED DESCRIPTION:
The aim of this study is to compare the clinical efficacy and the tolerance of assist control and pressure support modes during domiciliary noninvasive ventilation in patients with chronic respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Chronic respiratory failure
* Clinical symptoms of chronic alveolar hypoventilation
* PaCO2 ≥ 45 mmHg in case of restrictive pulmonary disorder or PaCO2 ≥ 55 mmHg in case or obstructive pulmonary disorder

Exclusion Criteria:

* Clinical exacerbation during the three previous weeks
* Previous treatment by domiciliary non invasive ventilation
* Previous treatment by non invasive ventilation for acute respiratory failure during the 3 previous months
* Bronchiectasis
* Duchenne muscular dystrophy
* Amyotrophic lateral sclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-01; Primary Completion 2009-06 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
PaO2 | months
  Blood gases response to ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Antoine CUVELIER, MD, PhD, Principal Investigator — University Hospital, Rouen